CLINICAL TRIAL: NCT00699972
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation, Parallel-Group Study to Evaluate the Efficacy and Safety of E2007 (Perampanel) Given as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Brief Title: Evaluating the Efficacy and Safety of E2007 (Perampanel) Given as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-G000-304
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2015-10

CONDITIONS: Refractory Partial Seizures
Keywords: E2007; perampanel; refractory partial seizures; adjunctive therapy; seizure frequency; partial onset seizures; reduction in seizure frequency; safety; concomitant AED(s)
MeSH Terms: conditions — Seizures | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: E2007 (perampanel)
- 2 (Experimental)
  Interventions: Drug: E2007 (perampanel)
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2007 (perampanel) — 8 mg perampanel in a 1:1:1 ratio, 125 subjects/arm. All subjects will take a maximum of 6 tablets daily for the duration of the study and will be up-titrated weekly in 2-mg increments to their randomized dose.
  Other Names: Perampanel
  Arms: 1
Drug: E2007 (perampanel) — 12 mg perampanel in a 1:1:1 ratio, 125 subjects/arm. All subjects will take a maximum of 6 tablets daily for the duration of the study and will be up-titrated weekly in 2-mg increments to their randomized dose.
  Other Names: Perampanel
  Arms: 2
Drug: Placebo — Placebo in a 1:1:1 ratio, 125 subjects/arm. All subjects will take a maximum of 6 tablets daily for the duration of the study.
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and tolerability of perampanel when given as an adjunctive therapy in subjects with refractory partial seizures.

ELIGIBILITY:
Inclusion criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Provide written informed consent signed by the subject or legal guardian prior to entering the study or undergoing any study procedures (If the written informed consent is provided by the legal guardian because the subject is unable to do so, a written or verbal assent from the subject must also be obtained).
2. Be considered reliable and willing to be available for the study period and able to record seizures and report Adverse Events (AEs) them self or have a caregiver who can record seizures and report AEs for them.
3. Male or female and greater than or equal to 12 years of age (within the course of the study).
4. Females should be either of non-childbearing potential (defined as having undergone surgical sterilization, or postmenopausal [age 50 and amenorrheic for 12 months]) or of childbearing potential. Females of childbearing potential must have a negative serum Beta Human Chorionic Gonadotropin (ß-hCG) at Visit 1 and a negative urine pregnancy test prior to randomization at Visit 2. Female subjects of childbearing potential must agree to be abstinent or to use at least 1 medically acceptable method of contraception (eg, a double-barrier method [eg, condom + spermicide, condom + diaphragm with spermicide], IUD, or have a vasectomised partner) starting at Visit 1 and throughout the entire study period and for 2 months after the last dose of study drug. Those women using hormonal contraceptives must also be using an additional approved method of contraception (as described previously) starting at Visit 1 and continuing throughout the entire study period and for 2 months after the last dose of study drug. (It is not required for male subjects to use contraceptive measures based on preclinical toxicology data).
5. Have a diagnosis of epilepsy with partial seizures with or without secondarily generalized seizures according to the International League Against Epilepsy's Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history and an electroencephalogram (EEG) that is consistent with localization-related epilepsy; normal interictal EEGs will be allowed provided that the subject meets the other diagnosis criterion (ie, clinical history).
6. Have had a computed tomography (CT) or magnetic resonance imaging (MRI) within the last 10 years that ruled out a progressive cause of epilepsy.
7. Have uncontrolled partial seizures despite having been treated with at least 2 different anti-epileptic drugs (AEDs) within approximately the last 2 years.
8. During the 6-week Pre-randomization Phase subjects must have had ≥5 partial seizures per 6-week (with ≥2 partial seizures per each of 3-week period) and with no 25-day seizure-free period in the 6-week period, as documented via a valid seizure diary. Only simple partial seizures with motor signs, complex partial seizures, and complex partial seizures with secondary generalization are counted toward this inclusion.
9. Are currently being treated with stable doses of 1, 2 or a maximum of 3 approved AEDs. Only 1 inducer AED (defined as; carbamazepine, phenytoin, phenobarbital, or primidone only) out of the maximum of 3 AEDs is allowed.
10. Are on a stable dose of the same concomitant AED(s) for 1 month (or no less than 21 days) prior to Visit 1; in the case where a new AED regime has been initiated for a subject, the dose must be stable for 2 months (or no less than 49 days) prior to Visit 1.
11. If on a stable dose (other than intermittent rescue use) of benzodiazepines for epilepsy (or for anxiety or sleep disorders) the prescribed dose must be stable for 1 month (or no less than 21 days) prior to Visit 1. (Note: the use of intermittent rescue benzodiazepines is defined in the exclusion criterion #22 below.) When used in these cases (epilepsy, anxiety or sleep disorders), benzodiazepines will be counted as 1 AED; therefore, only 1 or a maximum of 2 additional approved AEDs will be allowed.
12. A vagal nerve stimulator (VNS) is allowed but it must have been implanted ≥5 months prior to Visit 1. Stimulator parameters can not be changed for 1 month (or no less than 21 days) prior to Visit 1 or thereafter during the study.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Participated in a study involving administration of an investigational compound or device within 1 month (or no less than 21 days) prior to Visit 1, or within approximately 5 half-lives of the previous investigational compound, whichever is longer.
2. Pregnant and/or lactating.
3. Participated in previous perampanel studies.
4. Presence of nonmotor simple partial seizures only.
5. Presence of primary generalized epilepsies or seizures, such as absences and or myoclonic epilepsies.
6. Presence or previous history of Lennox-Gastaut syndrome.
7. A history of status epilepticus within approximately 12 months prior to Visit 1.
8. Seizure clusters where individual seizures cannot be counted.
9. A history of psychogenic seizures.
10. Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the Investigator(s) could affect the subject's safety or the study conduct.
11. Scheduled and/or confirmed to have epilepsy surgery within 6 months after Visit 1; however those who have previously documented "failed" epilepsy surgery will be allowed.
12. Evidence of significant active hepatic disease. Stable elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) due to concomitant medication(s) will be allowed if they are less than 3 times the upper limit of normal (ULN).
13. Evidence of significant active hematological disease; white blood cell (WBC) count <= 2500/µL (2.50 1E+09/L) or an absolute neutrophil count <= 1000/µL (1.00 1E+09/L).
14. A clinically significant electrocardiogram (ECG) abnormality, including prolonged QTc defined as >450 msec.
15. Suffering from psychotic disorder(s) and/or unstable recurrent affective disorder(s) evident by use of antipsychotics or have had a suicide attempt(s) within approximately the last 2 years.
16. Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
17. History of drug or alcohol dependency or abuse within approximately the last 2 years.
18. Have had multiple drug allergies or a severe drug reaction to an AED(s), including dermatological (eg, Stevens-Johnson syndrome), hematological, or organ toxicity reactions.
19. If felbamate is used as a concomitant AED, subjects must be on felbamate for at least 2 years, with a stable dose for 2 months (or no less than 49 days) prior to Visit 1. They must not have a history of white blood cell (WBC) count below 2500/µL (2.50 1E+09/L), platelets below 100,000, liver function tests (LFTs) above 3 times the upper limit of normal (ULN), or other indication of hepatic or bone marrow dysfunction while receiving felbamate. If subjects received felbamate in the past, it must have been discontinued 2 months (or no less than 49 days) prior to Visit 1.
20. Concomitant use of vigabatrin. Subjects who took vigabatrin in the past must be off vigabatrin for approximately 5 months prior to Visit 1 and must have documentation showing no evidence of a vigabatrin associated clinically significant abnormality in a visual perimetry test.
21. Concomitant use of barbiturates (except for seizure control indication) within 1 month (or no less than 21 days) prior to Visit 1.
22. Use of intermittent rescue benzodiazepines (ie, 1-2 doses over a 24-hr period considered one-time rescue) 2 or more times in a 1-month period prior to Visit 1; or
23. Any condition(s) that will make the subject, in the opinion of the Investigator, unsuitable for the study.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2008-04-30; Primary Completion 2010-10-19 (Actual); Study Completion 2010-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, M.D., Study Director — Eisai Inc.
Locations (96):
- United States (59):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital And Medical Center, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Bright Minds Institute, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Mile High Research Center, Denver, Colorado
  - Children's Research Institute, Washington D.C., District of Columbia
  - University of Florida Health Sciences, Jacksonville, Jacksonville, Florida
  - Pediatric Neurology and Epilepsy Center, Loxahatchee Groves, Florida
  - Loxahatchee Groves, Florida
  - Pediatric Neurology PA, Orlando, Florida
  - North West Florida Clinical Research Group, Pensacola, Florida
  - Child Neurology Center Of Nw Florida, Pensacola, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Ronald Aung-Din, MD, PC, Sarasota, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - PANDA, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Georgia Neurology and Sleep Medicine Associates, Suwanee, Georgia
  - Josephson Wallack Munshower Neurology, Indianapolis, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Via Christi Comprehensive Epilepsy Center, Wichita, Kansas
  - Wichita, Kansas
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Kentucky Neuroscience Research, Louisville, Kentucky
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Neurology/Johns Hopkins Hospital, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Michigan Neurology Associates, P.C., Clinton Township, Michigan
  - Washington University, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Five Towns Neurology, PC, Cedarhurst, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Univeristy of Rochester Strong Epilepsy Center, Rochester, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Children's Hospital Medical Center Of Akron D/B/A Akron Children's Hospital, Akron, Ohio
  - University Neurology, Inc., Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University Of Toledo Medical Center, Toledo, Ohio
  - Neurological Associates of Tulsa, Inc., Tulsa, Oklahoma
  - Providence St. Vincent's Epilepsy Center, Portland, Oregon
  - Blair Medical Assiciates, Inc., Altoona, Pennsylvania
  - Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Le Bonheur Pediatric Specialists, Memphis, Tennessee
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Neurological Clinic of Texas, P.A., Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Regional Epilepsy Center, Milwaukee, Wisconsin
- Argentina (12):
  - Sanatorio Allende, Córdoba, Córdoba Province
  - Hospital San Roque, Córdoba, Córdoba- Provincia de Córdoba
  - Hospital Santa Clara de Asis, Salta, Salta Province
  - FLENI (Fundación para la Lucha Contra Las Enfermedades Neurológicas de La Infancia), Capital Federal- Provincia de Buenos Aires
  - Hospital Británico, Capital Federal- Provincia de Buenos Aires
  - Hospital de Niños Ricardo Gutiérrez, Capital Federal- Provincia de Buenos Aires
  - Hospital General de Agudos José María Ramos Mejia, Capital Federal- Provincia de Buenos Aires
  - Hospital General de Agudos Teodoro Álvarez, Capital Federal- Provincia de Buenos Aires
  - Hospital Italiano de Buenos Aires, Capital Federal- Provincia de Buenos Aires
  - Policlínica Bancaria 9 de Julio, Capital Federal- Provincia de Buenos Aires
  - Centro de Estudio y Tratamiento de la Epilepsia y Sueño- CETES S.A., Córdoba
  - Sanatorio Parque, Rosario
- Brazil (11):
  - Faculdade de Ciências Médicas - UNICAMP, Campinas
  - Hospital de Clinicas da UFPR, Curitiba
  - Santa Casa de Porto Alegre, Porto Alegre
  - HC Ribeirão Preto, Ribeirão Preto
  - Hospital Pedro Ernesto - UERJ, Rio de Janeiro
  - Hospital Universitário Professor Edgar Santos, Salvador
  - Faculdade de Medicinade São José do Rio preto, São José do Rio Preto
  - HC-FMUSP, São Paulo
  - Hospital Brigadeiro, São Paulo
  - Hospital Santa Marcelina, São Paulo
  - UNIFESP, São Paulo
- Canada (5):
  - Foothills Medical Center, Calgary, Alberta
  - London Health Sciences Center, London, Ontario
  - Youthdale Treatment Centers, Toronto, Ontario
  - Neuro Rive-Sud, Greenfield Park, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
- Chile (4):
  - Hospital Barros Luco Trudeau, Santiago
  - Hospital Base Valdivia Servicio de Neurología, Santiago
  - Hospital Dr. Sótero del Río, Santiago
  - Neuropsicología Ltda., Santiago
- Mexico (5):
  - MIRC, Monterrey, Nuevo Leon CP
  - Instituto Biomedico de Investigacion AC, Aguascalientes
  - Sarug Reyes, Aguascalientes
  - Medica Sur SIF-BIOTEC, Mexico City
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City

REFERENCES:
- [Result] French JA, Krauss GL, Biton V, Squillacote D, Yang H, Laurenza A, Kumar D, Rogawski MA. Adjunctive perampanel for refractory partial-onset seizures: randomized phase III study 304. Neurology. 2012 Aug 7;79(6):589-96. doi: 10.1212/WNL.0b013e3182635735. Epub 2012 Jul 25. PMID 22843280
- [Derived] Bresnahan R, Hill RA, Wang J. Perampanel add-on for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD010961. doi: 10.1002/14651858.CD010961.pub2. PMID 37059702
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920
- [Derived] French JA, Gil-Nagel A, Malerba S, Kramer L, Kumar D, Bagiella E. Time to prerandomization monthly seizure count in perampanel trials: A novel epilepsy endpoint. Neurology. 2015 May 19;84(20):2014-20. doi: 10.1212/WNL.0000000000001585. Epub 2015 Apr 15. PMID 25878175
- [Derived] Rosenfeld W, Conry J, Lagae L, Rozentals G, Yang H, Fain R, Williams B, Kumar D, Zhu J, Laurenza A. Efficacy and safety of perampanel in adolescent patients with drug-resistant partial seizures in three double-blind, placebo-controlled, phase III randomized clinical studies and a combined extension study. Eur J Paediatr Neurol. 2015 Jul;19(4):435-45. doi: 10.1016/j.ejpn.2015.02.008. Epub 2015 Mar 5. PMID 25823975
- [Derived] Steinhoff BJ, Ben-Menachem E, Ryvlin P, Shorvon S, Kramer L, Satlin A, Squillacote D, Yang H, Zhu J, Laurenza A. Efficacy and safety of adjunctive perampanel for the treatment of refractory partial seizures: a pooled analysis of three phase III studies. Epilepsia. 2013 Aug;54(8):1481-9. doi: 10.1111/epi.12212. Epub 2013 May 10. PMID 23663001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 534 participants were screened for entry into the study. Of 534 participants, 147 were screen failures and 387 were eligible to continue in the study. A total of 390 participants were randomized into the study; 387 who were eligible and 3 who failed screening but were inappropriately randomized (2 received study treatment and 1 did not).
Pre-assignment Details: This was a randomized, double-blind, placebo-controlled study consisting of three phases: Prerandomization, Double-blind, and Follow-up. Participants who experienced the required minimum number of seizures during prerandomization, entered the Double-blind Phase and were randomized to placebo or 8 or 12 mg perampanel groups.
Groups:
- Placebo: 6 placebo tablets received daily during both Titration and Maintenance Periods.
- Perampanel 8mg: Perampanel 8mg maximum daily dose (Titration from 2mg to 8mg daily over 6-weeks; Maintenance at 8mg daily over 13-weeks)
- Perampanel 12mg: Perampanel 12mg maximum daily dose (Titration from 2mg to 12mg daily over 6-weeks; Maintenance at 12mg daily over 13-weeks)
Period: Overall Study
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Started | 122 | 133 | 135
Completed | 106 | 114 | 100
Not Completed | 16 | 19 | 35
Not completed — Adverse Event | 7 | 9 | 24
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 7 | 4
Not completed — Lack of Efficacy | 2 | 0 | 2
Not completed — Administrative/Other | 3 | 1 | 4
Not completed — Randomized, Not Treated | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg | Total
Number analyzed (Participants) | 121 | 133 | 134 | 388
Age, Customized [Number; unit: participants] — Safety Population used. One subject in Arm 1 and one subject in Arm 3 were randomized, but not treated.
  participants
    <18 years | 14 | 15 | 10 | 39
    18-64 years | 102 | 116 | 119 | 337
    >64 years | 5 | 2 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population used. One subject in Arm 1 and one subject in Arm 3 were randomized, but not treated.
  Participants
    Female | 67 | 68 | 65 | 200
    Male | 54 | 65 | 69 | 188
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Number; unit: participants] — Safety Population used. One subject in Arm 1 and one subject in Arm 3 were randomized, but not treated.
  participants
    White | 103 | 115 | 116 | 334
    Black or African American | 13 | 6 | 8 | 27
    Asian | 0 | 1 | 1 | 2
    Chinese | 0 | 1 | 1 | 2
    American Indian or Alaska Native | 0 | 4 | 2 | 6
    Other | 5 | 6 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the 28-day Seizure Frequency From Baseline to the End of the Double-blind Phase (Titration and Maintenance Phases)
Description: Seizure frequency per 28 days was derived from the information recorded in the subject diaries.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full Intent-to-Treat (ITT) Analysis Set included all participants who were randomized to study drug, received study drug, and had any seizure frequency data during the Double-blind Phase.
Measure: Median (Full Range); unit: Percent Change in seizure frequency
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Number analyzed (Participants) | 121 | 133 | 133
Percent Change in seizure frequency | -20.95 [-100.0 to 397.5] | -26.34 [-100.0 to 150.7] | -34.49 [-100.0 to 659.7]

2. Secondary Outcome: Percentage of Participants Who Were Responders
Description: A responder was a participant who had a 50 percent or greater reduction in seizure frequency per 28 days from the Pre-randomization phase.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full ITT Analysis Set; Last Observation Carried Forward (LOCF)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Number analyzed (Participants) | 121 | 133 | 133
Percentage of Participants
  Yes (Responder) | 26.4 | 37.6 | 36.1
  No (Non-Responder) | 73.6 | 62.4 | 63.9

3. Secondary Outcome: Percent Change in the 28-day Complex Partial Plus Secondarily Generalized Seizure Frequency From Baseline to the End of the Double-blind Phase (Titration and Maintenance Phases)
Description: Percent Change in the Seizure frequency per 28 days was derived from the information recorded in the subject diaries.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full ITT Analysis Set
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Number analyzed (Participants) | 110 | 120 | 120
Percent Change | -17.88 [-100.0 to 653.5] | -33.03 [-100.0 to 150.7] | -33.06 [-100.0 to 1006.5]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose of the study drug (up to Day 161)
Description: Adverse events (AE) were assessed at clinical visits based on the subject's diary, vitals, weight, physical exam, neurological exam, laboratory evaluations; and by telephone interviews/contact. Safety Population used which consists of subjects who were randomized to study drug, received study drug, and had at least one postdose safety assessment.
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/133 | 0/134
Serious Adverse Events (participants affected / at risk) | 6/121 | 8/133 | 9/134
Other Adverse Events (participants affected / at risk) | 71/121 | 101/133 | 98/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | Perampanel 8mg (N=133) | Perampanel 12mg (N=134)
Convulsion (Nervous system disorders) | 0 | 1 | 2
Grand mal convulsion (Nervous system disorders) | 1 | 1 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Impulse-control disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple drug overdose intentional (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 2 | 0
Omental infarction (Gastrointestinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Skin graft (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | Perampanel 8mg (N=133) | Perampanel 12mg (N=134)
Vertigo (Ear and labyrinth disorders) | 0 | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 9 | 6
Nausea (Gastrointestinal disorders) | 8 | 9 | 8
Vomiting (Gastrointestinal disorders) | 5 | 4 | 7
Fatigue (General disorders) | 5 | 10 | 11
Irritability (General disorders) | 6 | 10 | 19
Influenza (Infections and infestations) | 8 | 6 | 4
Nasopharyngitis (Infections and infestations) | 6 | 10 | 6
Fall (Injury, poisoning and procedural complications) | 8 | 13 | 17
Weight increased (Investigations) | 1 | 8 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 7
Ataxia (Nervous system disorders) | 0 | 8 | 16
Balance disorder (Nervous system disorders) | 1 | 10 | 5
Dizziness (Nervous system disorders) | 12 | 50 | 51
Headache (Nervous system disorders) | 16 | 20 | 18
Somnolence (Nervous system disorders) | 16 | 24 | 23
Anxiety (Psychiatric disorders) | 3 | 7 | 7
Insomnia (Psychiatric disorders) | 6 | 8 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 8
Convulsion (Nervous system disorders) | 2 | 7 | 4
Aggression (Psychiatric disorders) | 0 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other